CLINICAL TRIAL: NCT02760862
Title: Comparative Study Between Hydrocortisone and Mannitol in Treatment of Postdural Puncture Headache: a Randomized Double-blind Study
Brief Title: Comparative Study Between Hydrocortisone and Mannitol in Treatment of Postdural Puncture Headache
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dr.Ibrahim Mamdouh Esmat, Dr.Ibrahim Mamdouh Esmat, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1102
Record Dates: First submitted 2016-04-29; First posted 2016-05-04 (Estimated); Results first posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Headache
MeSH Terms: conditions — Headache | interventions — Hydrocortisone; Mannitol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Group (I) (N=25) (Active Comparator): Group (I), received hydrocortisone 100mg, dissolved in 2ml normal saline, intravenously/8 hours for 48 hours (Hydrocortisone as sodium succinate, vial, equivalent to hydrocortisone 100mg, Egyptian INT, Pharmaceutical Industries CO. ARE,EIPICO.EGYPT).
  Interventions: Drug: hydrocortisone 100mg.
- Group (II) (N=25) (Active Comparator): group (II), received mannitol 20% intravenous fluid (100ml intravenously which was given over 30 minutes and followed by 100 ml on a 12hour basis for 48 hours) (Manufactured by Allmed Middle East, Egypt).
  Interventions: Drug: mannitol 20% intravenous fluid

INTERVENTIONS:
Drug: hydrocortisone 100mg. — Group (I), received hydrocortisone 100mg, dissolved in 2ml normal saline, intravenously/8 hours for 48 hours
  Other Names: (Hydrocortisone as sodium succinate, vial, equivalent to hydrocortisone 100mg, Egyptian INT, Pharmaceutical Industries CO. ARE,EIPICO.EGYPT)
  Arms: Group (I) (N=25)
Drug: mannitol 20% intravenous fluid — group (II), received mannitol 20% 100ml intravenously which was given over 30 minutes and followed by 100 ml on a 12hour basis. Urinary catheter was inserted for patients in group (II) under complete aseptic conditions by the anesthesia resident before the start of mannitol infusion and removed after its discontinuation, accompanied by the intravenous fluid infusion over 48 hours of 500ml of normal saline or Ringer's solution every 8 hours and the input/output fluid chart for evaluation of fluid balance.
  Other Names: mannitol 20% (Manufactured by Allmed Middle East, Egypt).
  Arms: Group (II) (N=25)

SUMMARY:
Fifty patients of both sex, aged 18-50 years and ASA I and II undergoing elective lower abdominal and pelvic surgery under spinal anesthesia were included in this randomized double-blind study. Patients were randomly divided into 2 groups 25 each; group (I) received intravenous hydrocortisone 100mg every 8 hours for 48 hours and group (II) received intravenous infusion of mannitol 20% 100ml over 30 minutes followed by 100ml every 12hours. Mean (+/- SD) of headache intensity at 0, 6, 12, 24 and 48 hours after beginning of treatment was assessed using visual analog scale.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-50 years old.
* both sex.
* ASA physical status I and II.
* 70-90 kg body weight.
* height 160-180 cm.
* Elective lower abdominal and pelvic surgery e.g. repair of inguinal hernia, repair of incisional hernia, varicocele and hydrocele.

Exclusion Criteria:

* Patients with impaired kidney or liver functions.
* history of cardiac or central nervous system disease.
* uncontrolled medical disease (diabetes mellitus and hypertension)
* history of intake of non-steroidal anti-inflammatory drugs or opioids within 24 h before surgery
* allergy to the used medications
* patient's refusal
* duration of surgery more than 120 minutes.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group (I) (N=25) | Group (II) (N=25)
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group (I) (N=25) | Group (II) (N=25) | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (9.1) | 35.1 (7.7) | 35.4 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 15 | 14 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Egypt | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients (in Digits) Got Earlier Relief of PDPH (in Hours) After Use of Hydrocortisone or Mannitol.
Time Frame: within 48 hours after starting of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Group (I) (N=25) | Group (II) (N=25)
Number analyzed (Participants) | 25 | 25
Participants | 25 | 25

ADVERSE EVENTS:
Arm/Group | Group (I) (N=25) | Group (II) (N=25)
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 2/25 | 0/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group (I) (N=25) (N=25) | Group (II) (N=25) (N=25)
flushing (Skin and subcutaneous tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No